CLINICAL TRIAL: NCT01005290
Title: Cardiovascular Fixed Dose Combination Pill: A Pharmacodynamic Interaction Study to Evaluate the Effect of a Fixed Dose Combination of Acetylsalicylic Acid, Simvastatin and Ramipril (Cardiovascular Fixed Dose Combination Pill) on Blood Pressure
Brief Title: A Pharmacodynamic Study to Evaluate the Effect of a Fixed Dose Combination Pill on Blood Pressure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Ferrer Internacional S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: P-080646-01
Record Dates: First submitted 2009-10-22; First posted 2009-10-30 (Estimated); Results first posted 2012-07-26 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-06

CONDITIONS: Hypertension
Keywords: cardiovascular; fixed; dose; combination; pill; hypertension
MeSH Terms: conditions — Hypertension | interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Ramipril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination pill (Experimental): A once daily oral dose of the cardiovascular fixed dose combination pill (containing 100 mg acetylsalicylic acid, 40 mg simvastatin, and 5 mg ramipril) for one week followed by a once daily oral dose of the cardiovascular fixed dose combination pill (containing 100 mg acetylsalicylic acid, 40 mg simvastatin, and 10 mg ramipril) for 4 weeks.
  Interventions: Drug: Combination pill
- Ramipril (Active Comparator): A once daily oral dose of 5 mg ramipril for one week followed by a once daily oral dose of 10 mg ramipril for 4 weeks.
  Interventions: Drug: Ramipril

INTERVENTIONS:
Drug: Combination pill — A once daily oral dose of the cardiovascular fixed dose combination pill (containing 100 mg acetylsalicylic acid, 40 mg simvastatin, and 5 mg ramipril) for one week followed by a once daily oral dose of the cardiovascular fixed dose combination pill (containing 100 mg acetylsalicylic acid, 40 mg simvastatin, and 10 mg ramipril) for 4 weeks.
  Arms: Combination pill
Drug: Ramipril — A once daily oral dose of 5 mg ramipril for one week followed by a once daily oral dose of 10 mg ramipril for 4 weeks.
  Arms: Ramipril

SUMMARY:
The purpose of this study is to compare the effect on systolic pressure of the 3 drugs given together in the cardiovascular combination pill (acetylsalicylic acid, simvastatin, and ramipril) to the effect on systolic pressure of ramipril given alone.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be ≥18 years old
* Previously untreated systolic pressure result of ≥120<160 mmHg and diastolic pressure result of ≥80<100 mmHg

Exclusion Criteria:

* Subjects must not have previously received any anti-hypertensive medication
* must not have a systolic pressure <120 mmHg or ≥160 mmHg and diastolic pressure result of <80 mmHg or ≥100 mmHg
* must not have had a previous coronary artery bypass graft (CABG)
* must not have had a previous percutaneous transluminal coronary angioplasty (PTCA) with a drug-eluting stent
* must not have severe congestive heart failure (New York Heart Classification [NYHC] III-IV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valentin Fuster, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ninety-four subjects were screened for eligibility, participants met eligibility requirements and entered the run-in period
Pre-assignment Details: 52 subjects enrered the run-in period with ramipril 2.5 mg, 38 subjects were randomized. 20 subjects were randomized to Sequence Combination pill/ Ramipril and 18 subjects to sequence Ramipril /Combination pill.
Groups:
- Pre-randomization Run-In: Screening period with ramipril 2.5 mg once daily
- Combination Pill Then Ramipril: After randomization, in Period 1 participants received a once daily oral dose of the cardiovascular fixed dose combination pill (containing 100 mg acetylsalicylic acid, 40 mg simvastatin, and 5 mg ramipril) for one week followed by a once daily oral dose of the cardiovascular fixed dose combination pill (containing 100 mg acetylsalicylic acid, 40 mg simvastatin, and 10 mg ramipril) for 4 weeks; participants received no intervention during wash-out; in Period 2 participants received a once daily oral dose of 5 mg ramipril for one week followed by a once daily oral dose of 10 mg ramipril for 4 weeks
- Ramipril Then Combination Pill: After randomization, in Period 1 participants received a once daily oral dose of 5 mg ramipril for one week followed by a once daily oral dose of 10 mg ramipril for 4 weeks; participants received no intervention during wash-out; in Period 2 participants received a once daily oral dose of the cardiovascular fixed dose combination pill (containing 100 mg acetylsalicylic acid, 40 mg simvastatin, and 5 mg ramipril) for one week followed by a once daily oral dose of the cardiovascular fixed dose combination pill (containing 100 mg acetylsalicylic acid, 40 mg simvastatin, and 10 mg ramipril) for 4 weeks.
Period: Run-In
Arm/Group | Pre-randomization Run-In | Combination Pill Then Ramipril | Ramipril Then Combination Pill
Started | 52 | 0 | 0
Completed | 38 | 0 | 0
Not Completed | 14 | 0 | 0
Period: Period 1 (5 Weeks)
Arm/Group | Pre-randomization Run-In | Combination Pill Then Ramipril | Ramipril Then Combination Pill
Started | 0 | 20 | 18
Completed | 0 | 13 | 9
Not Completed | 0 | 7 | 9
Period: Washout Period (2 Weeks)
Arm/Group | Pre-randomization Run-In | Combination Pill Then Ramipril | Ramipril Then Combination Pill
Started | 0 | 13 | 9
Completed | 0 | 13 | 9
Not Completed | 0 | 0 | 0
Period: Period 2 (5 Weeks)
Arm/Group | Pre-randomization Run-In | Combination Pill Then Ramipril | Ramipril Then Combination Pill
Started | 0 | 13 | 9
Completed | 0 | 13 | 7
Not Completed | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Randomized Patiens: All patients who were randomized to both treatment sequences
Arm/Group | Randomized Patiens
Number analyzed (Participants) | 38
Age Continuous [Mean (Standard Deviation); unit: years] | 39.8 (11.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 29
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Difference in the Adjusted Mean 24-h Systolic Pressure Results (Using ABPM) Between the Basal and the Final Visit of Each Treatment Period.
Description: Difference in the adjusted mean 24-h systolic pressure results using ABPM (Ambulatory Blood Pressure Monitoring)in the PP population.
Time Frame: Days 7 and 36 of Period 1 and days 49 and 85 of Period 2
Population: The PP set included all randomized subjects who received at least one dose of IMP, had a baseline primary endpoint measurement, had at least one post baseline primary endpoint measurement, and who had no major protocol deviations. The PP set served as the primary analysis set for analysis of the primary endpoint.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Combination Pill: Difference in the adjusted mean 24-h systolic pressure results (using ABPM) between the basal and the final visit of each treatment period.
- Ramipril: Difference in the adjusted mean 24-h diastolic pressure results (using ABPM) between the basal and the final visit of each treatment period.
Arm/Group | Combination Pill | Ramipril
Number analyzed (Participants) | 17 | 17
mm Hg | -2.40 (8.726) | -4.40 (8.173)

2. Secondary Outcome: Difference in the Adjusted Mean 24-h Diastolic Pressure Results Between the Basal and the Final Visit of Each Treatment Period
Description: Difference in the Adjusted Mean 24-h Diastolic Pressure Results (Using ABPM) Between the Basal and the Final Visit of Each Treatment Period
Time Frame: Days 7 and 36 of Period 1 and days 49 and 85 of Period 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Combination Pill; Ramipril: Difference in the adjusted mean 24-h diastolic pressure results (using ABPM) between the basal and the final visit of each treatment period.
Arm/Group | Combination Pill | Ramipril
Number analyzed (Participants) | 17 | 17
mm Hg | -1.85 (6.714) | -2.88 (5.731)

ADVERSE EVENTS:
Time Frame: Participants were followed for the whole study duration, an average of 18 weeks.
Arm/Group | Combination Pill | Ramipril
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/31
Other Adverse Events (participants affected / at risk) | 3/29 | 1/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Pill (N=29) | Ramipril (N=31)
Headache (Nervous system disorders) | 3 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Communications and publication must be agreed between sponsor and PI